CLINICAL TRIAL: NCT02460861
Title: Intraoperational Prostate Loge Biopsies (iPROLOGX) After Radical Prostatovesiculectomy (RPVE) in Prostate Cancer (PCA) Patients for Molecular Tumor Marker Analysis
Brief Title: Intraoperational Prostate Loge Biopsies (iPROLOGX) After Radical Prostatovesiculectomy
Acronym: iPROLOGX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Magdeburg (Other)
Collaborators: St. Antonius Hospital Gronau (Other)
Responsible Party: Principal Investigator, Johann J. Wendler, MD, Dr. med., University of Magdeburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MD-URO-00021
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Molecular staging; GSTP1; Surgical margins; prostatovesiculectomy
MeSH Terms: conditions — Prostatic Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PCA Magdeburg (Active Comparator): Prostate cancer conducted for RPVE with curative Intention, biopsies of the prostatic fossa in Magdeburg
  Interventions: Procedure: biopsies of the prostatic fossa in Magdeburg; Procedure: RPVE
- Non-prostate cancer Magdeburg/Gronau (Active Comparator): Conducted for CE in Male with bladder cancer or other indication for cystectomy but without prostate cancer in Magdeburg or Gronau, biopsies of the prostatic fossa in Gronau
  Interventions: Procedure: biopsies of the prostatic fossa in Magdeburg; Procedure: CE; Procedure: biopsies of the prostatic fossa in gronau
- PCA Gronau (Active Comparator): Prostate cancer conducted for ETRARP with curative Intention, biopsies of the prostatic fossa
  Interventions: Procedure: ETRARP; Procedure: biopsies of the prostatic fossa in gronau

INTERVENTIONS:
Procedure: biopsies of the prostatic fossa in Magdeburg — intraoperative Open surgical biopsies of the prostatic fossa after prostatevesiculectomy in Magdeburg
  Other Names: surgical biopsies
  Arms: Non-prostate cancer Magdeburg/Gronau; PCA Magdeburg
Procedure: RPVE — Open Radical prostatovesiculectomy in Magdeburg
  Other Names: surgical prostatectomy
  Arms: PCA Magdeburg
Procedure: ETRARP — Robotassisted Radical prostatovesiculectomy in Gronau
  Other Names: surgical prostatectomy
  Arms: PCA Gronau
Procedure: CE — Open cystectomy in Magdeburg/Gronau
  Other Names: surgical cystoprostatectomy
  Arms: Non-prostate cancer Magdeburg/Gronau
Procedure: biopsies of the prostatic fossa in gronau — intraoperative endoscopic robotassisted biopsies of the prostatic fossa after prostatevesiculectomy in Gronau
  Other Names: surgical biopsies
  Arms: Non-prostate cancer Magdeburg/Gronau; PCA Gronau

SUMMARY:
This project is about the detection of occult tumor cells in surgical margins of radical prostatovesiculectomy by analysing the methylation status of Glutathione S-transferase P 1 (GSTP1). After gland excision specimens are obtained from 9 defined areas of the prostatic fossa. The biopsies are divided into two parts. One part used for histopathological analysis and the other part for moleculargenetic analysis. Results will be correlated e.g. with tumor stage, Gleason Score and prostate specific antigen (PSA).

The prostate-cancer-negative control group with bladder cancer.

DETAILED DESCRIPTION:
This project is about the detection of occult tumor cells in surgical margins of radical prostatovesiculectomy by analysing the methylation status of Glutathione S-transferase P 1 (GSTP1). After gland excision specimens are obtained from 9 defined areas of the prostatic fossa. The biopsies are divided into two parts. One part used for histopathological analysis and the other part for moleculargenetic analysis. Results will be correlated e.g. with tumor stage, Gleason Score and prostate specific antigen (PSA).

The prostate-cancer-negative control group with bladder cancer.

DNA ISOLATION

DNA from biopsies stored by -80°C was isolated by using innuPREP DNA mini Kit (Analytik Jena, Jena, Germany) following protocol 1 of the manufacturer's instructions. DNA was eluted with 50 µl elution buffer. Concentration and purity were analysed by using Nanodrop 2000.

DNA BISULFITE MODIFICATION

DNA was modified by using EpiTect Bisulfite Kit (QIAGEN, Hilden, Germany) according to manufacturer's instructions. Samples were eluted once with 20 µl elution buffer.

QUANTITATIVE METHYLATION SPECIFIC PCR

Methylation status of GSTP1 is analysed by quantitative methylation-specific PCR (Q-MSP) using StepOnePlus Real-Time PCR System and StepOne Software v2.1 from Applied Biosystems (Darmstadt, Germany). Q-MSP was performed in duplicate analysing genes Actin and GSTP1. The primers' and testing probes' sequences used to amplify and detect hypermethylated GSTP1 were: 5'-AgTTgCgCggCgATTTC (forward primer), 5'-gCCCCAATACTAAATCACgACg (reverse primer) and 5'-CggTCgACgTTCggggTgTAgCg (taqman probe), labelled with fluorescence dye FAM. The primers' and testing probes' sequences used to amplify and detect Actin were: 5'-TggTgATggAggAggTTTAgTAAgT (forward primer), 5'-AACCAATAAAACCTACTCCTCCCTTAA (reverse primer),5'-ACCACCACCCAACACACAATAACAAACACA (taqman probe), labelled with fluorescence dye VIC.

The Q-MSP was carried out at 50°C for 2 min., 95°C for 15 min. followed by 50 cycles of 95°C for 1s and 60°C for 1 min. As a positive control bisulfite-converted DNA of DU145 and LNCap were used. Blank reactions with destillated water, which replaced DNA, served as negative control (NTC).

ELIGIBILITY:
Criteria for patients with prostate adenocarcinoma:

Inclusion Criteria

* sex: male
* diagnosis: prostate adenocarcinoma
* treatment: radical prostatovesiculectomy
* period of treatment: 11/30/2011 - 10/15/2013

Exclusion Criteria

* sex: female
* diagnosis: no prostate adenocarcinoma
* treatment: no radical prostatovesiculectomy
* period of treament: before 11/30/2011 or after 10/15/2013

Criteria for prostate adenocarcinoma negative control group:

Inclusion Criteria

* sex: male
* diagnosis: urothelial carcinoma
* treatment: cysto-prostatectomy
* period of treament: 12/14/2011 - 02/18/2014

Exclusion Criteria

* sex: female
* diagnosis: incidental prostate adenocarcinoma
* treatment: no cysto-prostatectomy
* period of treatment: before 12/14/2011 or after 02/18/2014

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Methylation status of GSTP1 | 2 years
  Methylation status of GSTP1 is analysed by quantitative methylation-specific PCR (Q-MSP)
Histopathology of prostate fossa biopsies | 2 years
  Histopathology of prostate fossa biopsies (Prostata cancer positive or negative)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schostak, Prof.Dr.med., Study Chair — University of Magdeburg
Locations (2):
- Germany (2):
  - St. Antonius Hospital, Gronau, North Rhine-Westphalia
  - Department of Urology, University Clinic Otto von Guericke University Magdeburg, Magdeburg, Saxony-Anhalt